CLINICAL TRIAL: NCT00309842
Title: Transplantation of Unrelated Umbilical Cord Blood for Patients With Hematological Diseases With Cyclophosphamide/Fludarabine/Total Body Irradiation Myeloablative Preparative Regimen
Brief Title: Myeloablative Umbilical Cord Blood Transplantation in Hematological Diseases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005LS043; UMN-MT2005-10 (Other: Blood and Marrow Transplantation Program); UMN-0507M71475 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2006-03-29; First posted 2006-04-03 (Estimated); Results first posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphocytic Leukemia; Chronic Myelogenous Leukemia; Myelofibrosis; MDS; Refractory Anemia; Chronic Lymphocytic Leukemia; Prolymphocytic Leukemia; Non-Hodgkin's Lymphoma; Leukemia; Lymphoma; Multiple Myeloma; Myelodysplastic Syndromes
Keywords: blastic phase chronic myelogenous leukemia; primary myelofibrosis; chronic myelomonocytic leukemia; myelodysplastic syndromes; juvenile myelomonocytic leukemia; recurrent adult Burkitt lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent lymphoblastic lymphoma; recurrent childhood acute myeloid leukemia; recurrent childhood large cell lymphoma; recurrent follicular lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; refractory chronic lymphocytic leukemia; refractory multiple myeloma; chronic myelogenous leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; multiple myeloma; adult lymphoblastic lymphoma; refractory anemia with excess blasts; refractory anemia; Burkitt lymphoma; childhood large cell lymphoma; adult Burkitt lymphoma; mantle cell lymphoma; childhood lymphoblastic lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Primary Myelofibrosis; Anemia, Refractory; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Prolymphocytic; Lymphoma, Non-Hodgkin; Leukemia; Lymphoma; Multiple Myeloma; Myelodysplastic Syndromes; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myelomonocytic, Juvenile; Burkitt Lymphoma; Lymphoma, Large-Cell, Immunoblastic; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Anemia, Refractory, with Excess of Blasts; Lymphoma, Mantle-Cell | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Cyclophosphamide; Cyclosporine; fludarabine phosphate; Mycophenolic Acid; Cord Blood Stem Cell Transplantation; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Unrelated UCBT for Blood Cancers (Experimental): Patients undergoing unrelated umbilical cord blood transplantation (UCBT) for hematologic malignancies treated with myeloablative preparative regimen comprising fludarabine phosphate, mycophenolate mofetil, filgrastim, cyclophosphamide, cyclosporine and fractionated total-body irradiation.
  Interventions: Biological: filgrastim; Drug: cyclophosphamide; Drug: cyclosporine; Drug: fludarabine phosphate; Drug: mycophenolate mofetil; Procedure: umbilical cord blood transplantation; Radiation: total-body irradiation

INTERVENTIONS:
Biological: filgrastim — All patients will receive G-CSF 5 mcg/kg/day intravenously(IV) (dose rounded to vial size) based on the actual body weight IV beginning on day +1 after umbilical cord blood (UCB) infusion. G-CSF will be administered daily until the absolute neutrophil count (ANC) exceeds 2.5 x 10^9/L for three consecutive days.
  Other Names: G-CSF
Drug: cyclophosphamide — Cyclophosphamide to be administered with high volume fluid flush and mesna (MT(S) 9006) at 10:00am, or per institutional routine, on days-7 and -6 after fludarabine. Cyclophosphamide 60mg/kg/day intravenous (IV) x 2 days, total dose 120 mg/kg (days -7 and -6) Dosing is calculated based on Actual BodyWeight (ABW) unless ABW > 30 kg above Ideal BodyWeight (IBW), in which case the dose should be computed using adjusted body weight.
  Other Names: Cytoxan
Drug: cyclosporine — Patients will receive cyclosporine (CSA) therapy beginning on day -3 maintaining a level of > 200 ng/mL. For adults the initial dose will be 2.5 mg/kg intravenously (IV) over 2 hours every 12 hours. For children < 40 kg the initial dose will be 2.5 mg/kg IV over 2 hours every 8 hours.
  Other Names: CSA
Drug: fludarabine phosphate — Fludarabine 25 mg/m2/day intravenously (IV) x 3 days, total dose 75 mg/m2 (days -8 to -6);
  Other Names: Fludara
Drug: mycophenolate mofetil — All patients will begin mycophenolate mofetil (MMF) on day -3. Patients ≥ 40 kilograms will receive MMF at the dose of 3 grams/day divided into 2 or 3 doses (every 12 or 8 hours).
  Pediatric patient (<40 kilograms) will receive MMF at the dose of 15 mg/kg three times a day.
  Other Names: MMF
Procedure: umbilical cord blood transplantation — The product is infused via intravenous (IV) drip directly into the central line without a needle, pump or filter.
  Other Names: UCBT
Radiation: total-body irradiation — The recommended TBI is 165 cGy given twice daily for a total dose of 1320 cGy (days -4 to -1).
  Other Names: TBI

SUMMARY:
RATIONALE: Giving chemotherapy drugs, such as fludarabine and cyclophosphamide, and total-body irradiation before a donor umbilical cord blood stem cell transplant helps stop the growth of cancer cells and prepares the patient's bone marrow for the stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving cyclosporine and mycophenolate mofetil may stop this from happening.

PURPOSE: This phase II trial is studying how well giving fludarabine and cyclophosphamide together with total-body irradiation works in treating patients who are undergoing an umbilical cord blood transplant for hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 1-year survival of patients undergoing unrelated umbilical cord blood transplantation (UCBT) for hematologic malignancies treated with myeloablative preparative regimen comprising fludarabine, cyclophosphamide, and fractionated total-body irradiation.

Secondary

* Determine the incidence of transplant-related mortality at 6 months after UCBT.
* Evaluate the pattern of chimerism after double UCBT.
* Determine the incidence of neutrophil engraftment at day 42 after UCBT.
* Determine the incidence of platelet engraftment at 6 months after UCBT.
* Determine the incidence of grade II-IV and grade III-IV acute graft-versus-host disease (GVHD) at day 100 after UCBT.
* Determine the incidence of chronic GVHD at 1 year after UCBT.
* Determine the disease-free survival at 1 and 2 years after UCBT.
* Determine the incidence of relapse at 1 year after UCBT.

OUTLINE: This is a nonrandomized, open-label, multicenter study.

* Preparative Regimen: Patients receive fludarabine IV over 1 hour on days -8 to -6 and cyclophosphamide IV on days -7 and -6. Patients also undergo total-body irradiation twice daily on days -4 to -1.
* Umbilical Cord Blood Transplantation (UCBT): Patients undergo 1 or 2 units of UCBT on day 0. Patients receive filgrastim (G-CSF) IV once daily beginning on day 1 and continuing until blood counts recover.
* Graft-versus-host disease (GVHD) prophylaxis: Patients receive cyclosporine IV over 2 hours 2 or 3 times daily beginning on day -3 and continuing until day 100 followed by a taper until day 180. Patients also receive mycophenolate mofetil IV or orally 2 or 3 times a day beginning on day -3 and continuing until day 30 or 7 days after engraftment in the absence of acute GVHD.

After completion of study treatment, patients are followed periodically for at least 5 years.

PROJECTED ACCRUAL: A total of 150 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Acute myeloid leukemia (AML): high risk CR1 (as evidenced by preceding myelodysplastic syndrome [MDS], high risk cytogenetics, ≥ 2 cycles to obtain complete remission [CR], erythroblastic or megakaryocytic leukemia; CR2+. All patients must be in CR as defined by hematological recovery, AND <5% blasts by light microscopy within the bone marrow with a cellularity of ≥15%.
* Very high risk pediatric patients with AML. Patients <21 years, however, are eligible with (M2 marrow) with < or = 25% blasts in marrow after having failed one or more cycles of chemotherapy. This group of patients will be analyzed separately.
* Acute lymphocytic leukemia (ALL): high risk CR1 [t(9;22), t (1:19), t(4;11) or other MLL rearrangements] hypodiploidy, or IKZF1 abnormalities), DNA index < 0.81, > 1 cycle to obtain CR or presence minimal residual disease (MRD). Patients in CR2+ are eligible. All patients must be in CR as defined by hematological recovery, AND <5% blasts by light microscopy within the bone marrow with a cellularity of ≥15%.
* Very high risk pediatric patients with ALL. patients <21 years are also considered high risk CR1 if they had M2 or M3 marrow at day 42 from the initiation of induction or M3 marrow at the end of induction. They are eligible once they achieved a complete remission
* Chronic myelogenous leukemia (CML) excluding refractory blast crisis. To be eligible in first chronic phase (CP1) patient must have failed or be intolerant to imatinib mesylate.
* Plasma Cell leukemia after initial therapy, who achieved at least a partial remission
* Advanced myelofibrosis
* Myelodysplasia (MDS) IPSS Int-2 or High risk (i.e. RAEB, RAEBt) or refractory anemia with severe pancytopenia or high risk cytogenetics. Blasts must be < 10% by a representative bone marrow aspirate morphology.
* Chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL), marginal zone B-cell lymphoma or follicular lymphoma are eligible if there was disease progression/relapse within 12 of achieving a partial or complete remission. Patients who had remissions lasting > 12 months, are eligible after at least two prior therapies. Patients with bulky disease (nodal mass greater than 5 cm) should be considered for debulking chemotherapy before transplant.
* Lymphoplasmacytic lymphoma, mantle-cell lymphoma, prolymphocytic leukemia are eligible after initial therapy in CR1+ or PR1+.
* Large cell NHL > CR2/> PR2. Patients in CR2/PR2 with initial short remission (<6 months) are eligible.
* Lymphoblastic lymphoma, Burkitt's lymphoma, and other high-grade NHL after initial therapy if stage III/IV in CR1/PR1 or after progression if stage I/II < 1 year.
* Multiple myeloma beyond PR2. Patients with chromosome 13 abnormalities, first response lasting less than 6 months, or β-2 microglobulin > 3 mg/L, may be considered for this protocol after initial therapy.
* Recipients must have a Karnofsky score (adults) ≥ 80 % or Lansky score ≥ 50% (pediatrics), and proper organ function.

Exclusion Criteria

* Active infection at time of transplantation
* History of human immunodeficiency virus (HIV) infection
* Pregnant or breast feeding.
* Chemotherapy refractory large cell and high grade NHL
* If < or = 18 years old, prior myeloablative transplant within the last 6 months. If >18 years old prior myeloablative allotransplant or autologous transplant
* Extensive prior therapy including > 12 months alkylator therapy or > 6 months alkylator therapy with extensive radiation.
* Patients who have received Y-90 ibritumomab (Zevalin) or I-131 tostumomab (Bexxar), as part of their salvage therapy.

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 213 (Actual)
Dates: Start 2005-07-28 (Actual); Primary Completion 2019-07-29 (Actual); Study Completion 2019-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudio G. Brunstein, MD, PhD, Study Chair — Masonic Cancer Center, University of Minnesota
Locations (2):
- United States (2):
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Result] Verneris MR, Brunstein CG, Barker J, MacMillan ML, DeFor T, McKenna DH, Burke MJ, Blazar BR, Miller JS, McGlave PB, Weisdorf DJ, Wagner JE. Relapse risk after umbilical cord blood transplantation: enhanced graft-versus-leukemia effect in recipients of 2 units. Blood. 2009 Nov 5;114(19):4293-9. doi: 10.1182/blood-2009-05-220525. Epub 2009 Aug 25. PMID 19706886
- [Derived] MacMillan ML, Weisdorf DJ, Brunstein CG, Cao Q, DeFor TE, Verneris MR, Blazar BR, Wagner JE. Acute graft-versus-host disease after unrelated donor umbilical cord blood transplantation: analysis of risk factors. Blood. 2009 Mar 12;113(11):2410-5. doi: 10.1182/blood-2008-07-163238. Epub 2008 Nov 7. PMID 18997171

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Unrelated UCBT for Blood Cancers
Started | 213
Completed | 212
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Unrelated UCBT for Blood Cancers
Number analyzed (Participants) | 212
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 76
  Between 18 and 65 years | 136
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96
  Male | 116
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 199
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 13
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 12
  White | 162
  More than one race | 6
  Unknown or Not Reported | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were Alive at 1 Year Transplant Overall Survival
Description: Number of patients alive at 1 year after transplant.
Time Frame: at 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Unrelated UCBT for Blood Cancers
Number analyzed (Participants) | 212
Participants | 130

2. Secondary Outcome: Number of Participants Who Died Due to Transplant
Description: Determine the incidence of transplant-related mortality at 6 months after UCBT
Time Frame: At Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Unrelated UCBT for Blood Cancers
Number analyzed (Participants) | 212
Participants | 58

3. Secondary Outcome: Number of Participants With Platelet Engraftment
Description: Determine the incidence of platelet engraftment (platelet recovery >50,000/uL) at 6 months after UCBT.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Unrelated UCBT for Blood Cancers
Number analyzed (Participants) | 212
Participants | 159

4. Secondary Outcome: Number of Participants With Neutrophil Engraftment
Description: Determine the incidence of neutrophil engraftment at day 42 after UCBT Patients diagnosed with graft failure (failure of absolute neutrophil count ANC > 5 x 10^8/L of donor origin by day +42)
Time Frame: Day 42
Measure: Count of Participants; unit: Participants
Arm/Group | Unrelated UCBT for Blood Cancers
Number analyzed (Participants) | 212
Participants | 21

5. Secondary Outcome: Number of Participants With Acute Graft-Versus-Host Disease
Description: Determine the incidence of grade II-IV and grade III-IV acute graft-versus-host disease (GVHD) at day 100 after UCBT. Patients will be staged weekly between days 0 and 100 after transplantation using standard criteria following Przepiorka et al, 1995, Consensus Clinical Stage and Grade of Acute GVHD.
  Patients will be assigned an overall GVHD score based on extent of skin rash, volume of diarrhea and maximum bilirubin level.
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Unrelated UCBT for Blood Cancers
Number analyzed (Participants) | 212
Participants
  Grade II-IV | 106
  Grade III-IV | 49

6. Secondary Outcome: Number of Participants With Chronic Graft-Versus-Host Disease
Description: Determine the incidence of chronic GVHD at 1 year after UCBT. Patients will be staged weekly between days 0 and 100 after transplantation using standard criteria.
  Patients will be assigned an overall GVHD score based on extent of skin rash, volume of diarrhea and maximum bilirubin level.
Time Frame: Year 1
Measure: Count of Participants; unit: Participants
Arm/Group | Unrelated UCBT for Blood Cancers
Number analyzed (Participants) | 212
Participants | 39

7. Secondary Outcome: Percentage Chimerism on Day 21
Description: Chimerism studies will be performed on the bone marrow on days 21 and 100 and at 6 months, 1 year and 2 years. In cases of slow engraftment a bone marrow biopsy may be repeated on day +28.
Time Frame: Day 21
Measure: Mean (Standard Deviation); unit: percentage of donor cells
Arm/Group | Unrelated UCBT for Blood Cancers
Number analyzed (Participants) | 212
percentage of donor cells | 92.6 (14.9)

8. Secondary Outcome: Percentage Chimerism on Day 100
Description: as for outcome 7
Time Frame: Day 100
Measure: Mean (Standard Deviation); unit: percentage of donor cells
Arm/Group | Unrelated UCBT for Blood Cancers
Number analyzed (Participants) | 212
percentage of donor cells | 98.1 (8.5)

9. Secondary Outcome: Percentage Chimerism at 6 Months
Description: as for outcome 7
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: percentage of donor cells
Arm/Group | Unrelated UCBT for Blood Cancers
Number analyzed (Participants) | 212
percentage of donor cells | 98.1 (11.3)

10. Secondary Outcome: Percentage Chimerism at 1 Year
Description: as for outcome 7
Time Frame: 1 Year
Measure: Mean (Standard Deviation); unit: percentage of donor cells
Arm/Group | Unrelated UCBT for Blood Cancers
Number analyzed (Participants) | 212
percentage of donor cells | 99.1 (8.5)

11. Secondary Outcome: Percentage Chimerism at 2 Years
Description: as for outcome 7
Time Frame: 2 Years
Measure: Mean (Standard Deviation); unit: percentage of donor cells
Arm/Group | Unrelated UCBT for Blood Cancers
Number analyzed (Participants) | 212
percentage of donor cells | 100 (0.1)

ADVERSE EVENTS:
Time Frame: Upto 2 years
Arm/Group | Unrelated UCBT for Blood Cancers
All-Cause Mortality (participants affected / at risk) | 161/212
Serious Adverse Events (participants affected / at risk) | 92/212
Other Adverse Events (participants affected / at risk) | 187/212
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Unrelated UCBT for Blood Cancers (N=212)
Acute respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 4 (4)
cardiopulmonary arrest (Cardiac disorders) | 1 (1)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 41 (41)
Graft failure (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9)
Graft versus host disease (GVHD) (Immune system disorders) | 13 (13)
Infection (Infections and infestations) | 10 (11)
Progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pulmonary hemorrage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary other (Respiratory, thoracic and mediastinal disorders) | 3 (3)
relapse (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Veno-Occlusive Disease (VOD) (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Unrelated UCBT for Blood Cancers (N=212)
Multi organ failure (General disorders) | 12 (13)
Hemorrhage (Blood and lymphatic system disorders) | 12 (14)
Neurotoxicity (Nervous system disorders) | 13 (14)
Neuropathy (Nervous system disorders) | 16 (16)
Acute kidney injury (Renal and urinary disorders) | 18 (18)
GI bleeding (Gastrointestinal disorders) | 18 (19)
Hypertension (Vascular disorders) | 62 (62)
Veno-Occlusive Disease (VOD) (Hepatobiliary disorders) | 12 (19)
Hyperglycemia (Metabolism and nutrition disorders) | 22 (22)
Dialysis (Renal and urinary disorders) | 23 (23)
Engraftment syndrome (General disorders) | 25 (25)
Acute respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 26 (27)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 34 (42)
Pericardial effusion (Cardiac disorders) | 46 (52)
Intubation (Respiratory, thoracic and mediastinal disorders) | 58 (74)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 131 (297)
Infection (Infections and infestations) | 126 (527)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-02-06): https://cdn.clinicaltrials.gov/large-docs/42/NCT00309842/Prot_SAP_000.pdf